CLINICAL TRIAL: NCT04117685
Title: A Prospective, Global Hip Dysplasia Registry with Follow-up to Skeletal Maturity: an Analysis of Risk Factors, Screening Practices and Treatment Outcomes
Brief Title: Global Hip Dysplasia Registry
Acronym: GHDR
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kishore Mulpuri, Professor, University of British Columbia
Other Study IDs: H16-01794
Record Dates: First submitted 2019-10-02; First posted 2019-10-07 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Hip Dislocation, Congenital; Hip Dysplasia, Congenital, Nonsyndromic; Congenital Dysplasia of the Hip; Congenital Hip Dislocation; Congenital Hip Displacement; Congenital Hip Dysplasia; Dislocation of Hip, Congenital; Dislocation, Congenital Hip; Displacement, Congenital Hip; Dysplasia, Congenital Hip; Hip Displacement, Congenital; Hip, Dislocation Of, Congenital
Keywords: hip dysplasia; ddh; developmental dysplasia of the hip; congenital hip dysplasia
MeSH Terms: conditions — Hip Dislocation, Congenital; Hip Dislocation; Developmental Dysplasia of the Hip | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Arm I: Prospective from diagnosis: Patients have been enrolled and followed since diagnosis will be placed into Arm I.
  Interventions: Other: Observational
- Arm II: Prior treatment at center: Patients who have received previous treatment and will continue to receive treatment at the participating center will be placed into Arm II.
  Interventions: Other: Observational
- Arm III: Prior treatment at outside center: Patients who have received previous treatment at an outside center but are continuing treatment at a participating center will be placed into Arm III.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — All groups will undergo observational data collection. No interventions will be made to patient care.

SUMMARY:
Developmental dysplasia of the hip (DDH) is the most common hip condition affecting infants and children. DDH represents a spectrum of issues affecting the hip joint - a "ball-and-socket" joint. When the femoral head (the "ball) is seated properly in the acetabulum (the "socket"), the hip is stable and can develop normally. However, when the femoral head is not well-seated, the hip can become unstable or dislocate. This instability or dislocation of the femoral head prevents the hip joint from developing normally during infancy and early childhood. If left undetected or untreated, it can lead to debilitating complications later in life.

Development of a comprehensive, prospective international registry for all infants and children with DDH will provide the potential to impact all infants born, not only in British Columbia, but around the world. The purpose of this initiative is to identify best practices and standardize treatment and management strategies in order to optimize clinical and functional outcomes for patients with DDH. This registry includes targeted specific outcomes that will be investigated, in addition to the general collection of data on all patients diagnosed with any form of DDH up to the age of 10 years.

DETAILED DESCRIPTION:
DDH is the most common pediatric hip condition, with 1-3% of all newborns diagnosed at birth. However, the true incidence of DDH is difficult to quantify due to significant variations in diagnostic criteria, terminology, screening and monitoring procedures, as well as ethnic and cultural differences. The spectrum of DDH encompasses mild dysplasia or instability of a reduced hip, to a completely dislocated, irreducible hip. If left undetected or untreated, it can lead to debilitating complications later in life. Much of the evidence existing to date in the DDH literature is from retrospective and/or single-centre studies, and the spectral nature of the condition has resulted in inconsistent or ill-defined terminology to classify patients in regard to diagnosis and laterality. Consequently, the patient population is often not clearly defined or reported, making it difficult to compare or combine different study results in order to produce strong evidence to guide treatment and management. This issue was highlighted in the updated clinical practice guidelines released in partnership between the American Academy of Orthopaedic Surgery (AAOS) and the Pediatric Orthopaedic Society of North America (POSNA) in 2014. Of the nine recommendations made, only two were of moderate strength, while the other seven were of low strength.

Discrepancies begin with DDH screening practices. Clinical examination for hip instability is a universal standard practice; however, not all cases are detectable by this method, leading to potential missed diagnoses or late-presentations that are more difficult to treat. Beyond the clinical exam, screening, management and treatment practices are highly variable across surgeons, centres and countries. Some countries, particularly those in Europe, employ universal ultrasound screening, while others use selective ultrasound screening as a supplement to the clinical exam for infants with specific risk factors. Defined risk factors that have currently been deemed to warrant further screening and monitoring include breech presentation, family history of DDH or a clinical history of hip instability. Regardless of screening program, missed or late-presentations still occur, warranting further investigation. Further variability is introduced with primary treatment and management. Bracing is the most common first-line treatment, particularly in younger patients or patients with unstable or reducible hips. Surgical treatment (closed or open reduction) is more often used as first-line treatment in older patients, or patients with more severe dislocations. However, significant variation is seen in practice patterns, complication rates and treatment success with each of these methods, and identification and analysis of prognostic factors have been lacking methodological rigor. Development of a comprehensive, prospective registry will provide a unique and unprecedented platform for examining numerous aspects of the full DDH spectrum, including long-term treatment outcomes and risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 0 and 10 years at time of initial diagnosis
* Referred for DDH screening due to specific risk factors OR diagnosed with DDH
* Diagnosis confirmed with appropriate ultrasonographic or radiographic imaging

Exclusion Criteria:

* Known or suspected neuromuscular, collagen, chromosomal or lower extremity congenital anomalies
* Teratologic hip dislocation (syndromic-associated dislocations)
* Over 10 years of age at initial diagnosis
* Received prior treatment for DDH without appropriate imaging or documentation

Ages: 1 Minute to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who have been referred to a participating center for DDH risk factors or patients with diagnosed DDH will be included in the registry. Patients will be enrolled during one of their routine clinic appointments at one of the participating centers.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of a general, prospective DDH registry with follow-up to skeletal maturity | Until study completion in 2028
  Data will be collected from patients with or at risk of DDH to create a registry. Patients will be followed up until skeletal maturity.
Identification of variation in DDH screening, diagnosis, and management protocols | Until study completion in 2028
  Using data from the registry, variation in DDH screening, diagnosis, and management protocols will be identified.
Comparison of brace treatment outcomes within and across diagnostic categories | Until study completion in 2028
  Using data from the registry, brace treatment outcomes within and across diagnostic categories will be compared.
Comparison of surgical treatment outcomes within and across diagnostic categories | Until study completion in 2028
  Using data from the registry, surgical treatment outcomes within and across diagnostic categories will be compared.
Identification of optimal timing of both bracing and surgical treatment | Until study completion in 2028
  Using data from the registry, optimal timing of both bracing and surgical treatment will be identified.
Identification and characterization of risk factors for treatment complications (i.e., AVN) | Until study completion in 2028
  Using data from the registry, risk factors for treatment complications (i.e., AVN) will be identified and characterized.
Identification of predictors of the need for hip reconstructive surgery in adolescence | Until study completion in 2028
  Using data from the registry, predictors of the need for hip reconstructive surgery in adolescence will be identified.

SECONDARY OUTCOMES:
Development of targeted sub-studies within the registry | Until study completion in 2028
  Using data from the registry, further targeted DDH sub-studies will be developed.
Assessment and analysis of risk factor screening and monitoring protocols for DDH by a non-inferiority randomized controlled trial (RCT) | Until study completion in 2028
  Risk factor screening and monitoring protocols for DDH by a non-inferiority RCT will be assessed and analyzed.
A comparison of rigid versus dynamic bracing in early treatment of DDH by RCT | Until study completion in 2028
  Rigid versus dynamic bracing in early treatment DDH by RCT will be compared.
A comparison of observation versus bracing in clinically stable, ultrasonographically dysplastic hips by RCT | Until study completion in 2028
  Observation versus bracing in clinically stable, ultrasonographically dysplastic hips by RCT will be compared.
An analysis of the impact of brace treatment length after hip stabilization by RCT | Until study completion in 2028
  The impact of brace treatment length after hip stabilization by RCT will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Mulpuri, FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No